CLINICAL TRIAL: NCT05219942
Title: Outcome of Using Long Acting Glargine Insulin With Low Dose Regular Insulin Infusion in Diabetic Ketoacidosis Patients :A Comparative Study
Brief Title: Outcome of Glargine Insulin in Renal Impairment Patients With Diabetic Ketoacidosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona Ammar, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R 103/ 2020
Record Dates: First submitted 2022-01-09; First posted 2022-02-02 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Insulin Glargine; Insulin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients of both groups know that they will receive crystalline insulin infusion.However they are not told whether they receive glargine insulin or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low dose insulin infusion +Subcutaneous saline (Placebo Comparator): low dose insulin infusion +Subcutaneous saline
  Interventions: Other: normal saline
- low dose insulin infusion +subcutaneous Glargine insulin (Active Comparator): low dose insulin infusion +subcutaneous Glargine insulin
  Interventions: Drug: Glargine

INTERVENTIONS:
Drug: Glargine — regular low dose insulin infusion 0.1 IU/Kg/hour and subcutaneous Glargine insulin (made by Sanofi®) within the first 2 hours of ICU admission. The dose of insulin glargine will be adjusted according to the calculated (eGFR > 90 dose = 0.27 IU/kg/day, eGFR 60-89 dose = 0.25 IU/kg/day, eGFR <60 dose = 0.19 IU/kg/day.
  Other Names: insulin
  Arms: low dose insulin infusion +subcutaneous Glargine insulin
Other: normal saline — regular low dose insulin infusion 0.1 IU/Kg/hour and subcutaneous saline instead of insulin glargine will be given in the control group.
  Arms: low dose insulin infusion +Subcutaneous saline

SUMMARY:
The study aims to compare between the use of continuous low dose insulin infusion versus co-administration of low dose continuous insulin infusion and early subcutaneous insulin glargine in diabetic ketoacidosis patients with chronic renal impairment. aim to investigate the effect of using the long acting insulin analogue glargine on the resolution time of diabetic ketoacidosis in renal impairment patients who have altered insulin pharmacokinetics and pharmacodynamics and the rate of adverse effects of this approach

DETAILED DESCRIPTION:
Diabetic ketoacidosis (DKA) is one of the most common and grave acute complications of diabetes and is a significant cause of morbidity and mortality.

The current available guidelines state that the most effective means of insulin delivery during DKA is a continuous low dose infusion of regular insulin. The patients must be admitted to the ICU for frequent and close monitoring .In addition to insulin infusion, correction of dehydration, and electrolyte and acid base disorders is achieved together with identification and treatment of co-morbid precipitating factors .

"The Joint British Diabetes Societies guideline for the management of diabetic ketoacidosis" recommends continuation of a long-acting insulin analogue such as insulin glargine during the initial management of DKA because it provides background insulin when the intravenous insulin is discontinue.

Administering basal insulin concomitantly with regular insulin infusion was found to be well tolerated, associated with faster resolution of acidosis without any adverse effects; patients required a shorter duration of intravenous insulin infusion and had a lower total dose of intravenous insulin and significantly decreased hyperglycemia after discontinuation of the intravenous insulin .

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients.
* Type I and type II diabetes mellitus.
* Patients on insulin and/or oral hypoglycemic therapy.
* Duration of diabetes more than 5 years.
* Medical and surgical patients.

Exclusion Criteria:

* Severe persistent hypotension (SBP <80 inspite of receiving 1000ml of normal saline).
* Acute myocardial infarction.
* Progressive renal failure or end stage renal disease defined as eGFR < 15ml/min.
* Liver cell failure.
* Pregnancy.
* Need for emergency surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Mean time to reversal of diabetic ketoacidosis | 48 hours
  Resolution of DKA is defined as blood sugar <200mg/dl plus any two of serum bicarbonate ≥15,pH>7.3, and anion gap less than or equal to 12
Total crystalline insulin consumption | 48 hours
  Total number of units of insulin infusion consumed for diabetic ketocidosis to resolve

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barski L, Kezerle L, Zeller L, Zektser M, Jotkowitz A. New approaches to the use of insulin in patients with diabetic ketoacidosis. Eur J Intern Med. 2013 Apr;24(3):213-6. doi: 10.1016/j.ejim.2013.01.014. Epub 2013 Feb 8. PMID 23395363
- [Background] Barski L, Brandstaetter E, Sagy I, Jotkowitz A. Basal insulin for the management of diabetic ketoacidosis. Eur J Intern Med. 2018 Jan;47:14-16. doi: 10.1016/j.ejim.2017.08.025. Epub 2017 Aug 31. PMID 28864157
- [Background] Chapter 1: Definition and classification of CKD. Kidney Int Suppl (2011). 2013 Jan;3(1):19-62. doi: 10.1038/kisup.2012.64. No abstract available. PMID 25018975
- [Background] Savage MW, Dhatariya KK, Kilvert A, Rayman G, Rees JA, Courtney CH, Hilton L, Dyer PH, Hamersley MS; Joint British Diabetes Societies. Joint British Diabetes Societies guideline for the management of diabetic ketoacidosis. Diabet Med. 2011 May;28(5):508-15. doi: 10.1111/j.1464-5491.2011.03246.x. PMID 21255074
- [Background] Svensson M, Yu ZW, Eriksson JW. A small reduction in glomerular filtration is accompanied by insulin resistance in type I diabetes patients with diabetic nephrophathy. Eur J Clin Invest. 2002 Feb;32(2):100-9. doi: 10.1046/j.1365-2362.2002.00949.x. PMID 11895456